CLINICAL TRIAL: NCT06572449
Title: A Phase 3b, Open-label, Multicenter, Two-Period, Slow-titration and Food Effect Study to Assess the Safety and Efficacy of KarXT in Participants With DSM-5 Schizophrenia
Brief Title: Study to Assess Safety and Effectiveness of Slowly Increasing Dose and Food Effect of KarXT in Participants With Schizophrenia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Karuna Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CN012-0048
Record Dates: First submitted 2024-08-08; First posted 2024-08-27 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-03

CONDITIONS: Schizophrenia
Keywords: BMS-986510; KarXT; DSM-5 Schizophrenia; Diagnostic and Statistical Manual of Mental Disorders; Mental Disorders
MeSH Terms: conditions — Schizophrenia; Disease; Mental Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- KarXT on empty stomach and with food (Experimental)
  Interventions: Drug: KarXT

INTERVENTIONS:
Drug: KarXT — Specified dose on specified days
  Other Names: BMS-986510

SUMMARY:
The purpose of this study is to assess the safety and efficacy of slowly increasing dose and food effect of KarXT in adult participants with schizophrenia.

ELIGIBILITY:
Inclusion Criteria:

* Has a primary diagnosis of schizophrenia established by a comprehensive psychiatric evaluation based on the DSM-5 (American Psychiatric Association 2013) criteria and confirmed by Mini International Neuropsychiatric Interview (MINI) for Schizophrenia and Psychotic Disorder Studies version 7.0.2.
* Positive and Negative Syndrome Scale (PANSS) total score of ≤ 80 at screening and Baseline.
* Clinical Global Impression-Severity (CGI-S) score of ≤ 4 at screening and Baseline.
* Willing and able to discontinue all antipsychotic medications prior to baseline visit.

Exclusion Criteria:

* History or presence of clinically significant cardiovascular, pulmonary, renal, hematologic, gastrointestinal (GI), endocrine, immunologic, dermatologic, neurologic, or oncologic disease or any other condition that, in the opinion of the investigator, would jeopardize the safety of the participant or the validity of the study results.
* Any primary DSM-5 disorder other than schizophrenia within 12 months before screening.
* History of treatment resistance to schizophrenia medications.
* History of allergy/hypersensitivity to KarXT.
* Other protocol-defined Inclusion/Exclusion criteria apply.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 173 (Actual)
Dates: Start 2024-10-28 (Actual); Primary Completion 2025-03-13 (Actual); Study Completion 2025-03-13 (Actual)

PRIMARY OUTCOMES:
Incidence of treatment-emergent adverse events (TEAEs) | Up to approximately 11 weeks

SECONDARY OUTCOMES:
Incidence of TEAEs by study period | Up to approximately 11 weeks
Incidence of serious TEAEs | Up to approximately 11 weeks
Incidence of serious TEAEs by study period | Up to approximately 11 weeks
Incidence of TEAEs leading to study intervention discontinuation | Up to approximately 11 weeks
Incidence of TEAEs leading to study intervention discontinuation by study period | Up to approximately 11 weeks
Incidence of pro- and anticholinergic TEAEs | Up to approximately 11 weeks
Incidence of pro- and anticholinergic TEAEs by study period | Up to approximately 11 weeks
Change from baseline in Positive and Negative Syndrome Scale (PANSS) total score | Up to approximately 11 weeks
Change from baseline in PANSS positive score | Up to approximately 11 weeks
Change from baseline in PANSS negative score | Up to approximately 11 weeks
Change from baseline in PANSS negative Marder Factor score | Up to approximately 11 weeks
Change from baseline in Clinical Global Impression-Severity (CGI-S) score | Up to approximately 11 weeks
Spontaneously reported adverse event of special interest (AESIs) | Up to approximately 11 weeks
Change from baseline in body weight | Up to approximately 11 weeks
Change from baseline in body mass index (BMI) | Up to approximately 11 weeks
Change from baseline in waist circumference | Up to approximately 11 weeks
Change from baseline in orthostatic vital signs (supine and standing after 2 minutes) at Day 7 and Day 14: blood pressure (systolic and diastolic) and heart rate | Up to approximately 11 weeks
  BP includes systolic and diastolic measurements (mm Hg); Heart rate is measured in beats/minute (bpm)
Change from baseline in blood pressure | Up to approximately 11 weeks
Change from baseline in heart rate | Up to approximately 11 weeks
Change from baseline in clinical laboratory assessment (Hematology) | Up to approximately 11 weeks
  Hematology will include full, differential blood [red blood cell (RBC), white blood cell (WBC)] and platelet counts, hemoglobin, hematocrit, mean corpuscular measures.
Change from baseline in clinical laboratory assessment (Clinical chemistry) | Up to approximately 11 weeks
  Clinical chemistry will include liver and kidney function tests along with metabolic, lipids panel and electrolytes.
Change from baseline in clinical laboratory assessment (Urinalysis) | Up to approximately 11 weeks
Change from baseline in clinical laboratory assessment (Drug screen) | Up to approximately 11 weeks
Change from baseline in 12-lead ECG [Ventricular rate (bpm)] | Up to approximately 11 weeks
Change from baseline in 12-lead ECG [PR interval (msec)] | Up to approximately 11 weeks
Change from baseline in 12-lead ECG [QRS interval (msec)] | Up to approximately 11 weeks
Change from baseline in 12-lead ECG [QT interval (msec)] | Up to approximately 11 weeks
Change from baseline in 12-lead ECG [QTcF interval (msec)] | Up to approximately 11 weeks
Change from baseline in physical examination | Up to approximately 11 weeks
  A complete (body temperature, general appearance, head/eyes/ears/nose/throat, examination of thorax and abdomen, assessment of cardiac, musculoskeletal, and circulatory systems, palpations for lymphadenopathy, and limited neurological examination) and targeted organ systems physical examinations will be performed.
Suicidal ideation scale with the use of Columbia-Suicide Severity Rating Scale (C-SSRS) | Up to approximately 11 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (6):
- United States (6):
  - Local Institution - 0002, Los Alamitos, California
  - Local Institution - 0004, Riverside, California
  - Local Institution - 0006, Hollywood, Florida
  - Local Institution - 0005, Atlanta, Georgia
  - Local Institution - 0003, Decatur, Georgia
  - Local Institution - 0001, Marlton, New Jersey

IPD SHARING:
Plan to Share IPD: Yes
BMS will provide access to individual anonymized participant data upon request from qualified researchers, and subject to certain criteria.
  Additional information regarding Bristol Myer Squibb's data sharing policy and process can be found at:
  https://www.bms.com/researchers-and-partners/clinical-trials-and-research/disclosurecommitment.html
Supporting Information: Study Protocol, SAP, CSR
Time Frame: See Plan Description
Access Criteria: See Plan Description
URL: https://www.bms.com/researchers-and-partners/clinical-trials-and-research/disclosure-commitment.html

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.BMSClinicalTrials.com